CLINICAL TRIAL: NCT04698408
Title: Dietary Intervention Trial Targeting Metabolic Syndrome After Renal Transplantation
Brief Title: Dietary Intervention Trial Targeting Metabolic Syndrome After Kidney Transplantation
Acronym: DIETTX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Stephan J.L. Bakker, prof. dr., University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: METc2020/050
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Kidney Transplant; Complications
Keywords: kidney transplantation; metabolic syndrome; high-protein diet; dietary intervention
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-protein, carbohydrate-reduced diet (Experimental)
  Interventions: Other: high-protein, carbohydrate-reduced diet
- Dutch Nutritional Guidelines (Active Comparator)
  Interventions: Other: Dutch Nutritional Guidelines

INTERVENTIONS:
Other: high-protein, carbohydrate-reduced diet — the high-protein, carbohydrate-reduced diet will consist of 1.2-1.4 g/kg/d protein, 26-20en% carbohydrates and +/- 50en% fatty acids, with mainly unsaturated fatty acids. This diet consist of mainly unprocessed, fresh nutrient-dense food-products. Ultra-processed foods and alcoholic beverages will be totally avoided. Salt consumption will not exceed 5-6 g/d. The diet is ad libitum and caloric restriction will not be applied. The diet will be followed for 6 weeks.
  Arms: high-protein, carbohydrate-reduced diet
Other: Dutch Nutritional Guidelines — the diet according to the Dutch Nutritional Guidelines will consist of a protein intake of 0.8-1.0 g/kg/d and 50-60en% carbohydrates, and +/-30en% fatty acids, with restriction of saturated fatty acids <10en%. This diet consist of mainly unprocessed, fresh nutrient-dense food-products. Ultra-processed foods and alcoholic beverages will be totally avoided. Salt consumption will not exceed 5-6 g/d. The diet is ad libitum and caloric restriction will not be applied. The diet will be followed for 6 weeks.
  Arms: Dutch Nutritional Guidelines

SUMMARY:
Kidney transplant recipients (KTR) have a considerably lower life expectancy as compared with the general population, primarily due to a high prevalence of cardiovascular diseases. KTR often develop an unfavourable cardio-metabolic risk profile characterized by weight gain, metabolic syndrome and post-transplantation diabetes mellitus (PTDM). In general, nutrition plays a key role in both the prevention and treatment of these cardio-metabolic derangements.

However, in KTR most RCT's with a dietary intervention, failed to show significant improvement in cardio-metabolic health. This at least questions the efficacy of the diets of these intervention, which relied on general or diabetes guidelines, after kidney transplantation. KTR not only face a high cardio-metabolic risk, but also have a high risk for malnutrition and muscle mass depletion. More knowledge is required to determine the optimal diet and macronutrient composition for improvement of the cardio-metabolic risk factors in the context of the high malnutrition risk. In this regard, observational studies point towards the needs for a higher protein intake for better patient outcomes. Therefore, in this study, the investigators will examine if a high-protein, carbohydrate-reduced diet is more effective than a diet in line with the Dutch Dietary Guidelines for improvement of cardio-metabolic risk factors and for improvement of the body composition in KTR.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Given informed consent.
* At least 6 months after kidney transplantation.
* Stable renal function with an estimated glomerular filtration rate (eGFR) > 30 mL/min.
* Raised systolic blood pressure (≥130 mmHg) and at least two more features of metabolic syndrome: central obesity (waist circumference ≥102 for men and ≥88cm for women), elevated triglycerides (≥ 1.7 mmol/L), reduced HDL-C (< 1.0 mmol/L for men and < 1.3 mmol/L for women) or on drug treatment for reduced HDL, elevated plasma glucose (≥ 5.6 mmol/L) or on drug treatment for elevated glucose9.
* Approval by nephrologist for participation in the study.

Exclusion Criteria:

* Active medical illness, including rejection of the graft.
* Psychopathology or serious cognitive impairment.
* Necessity to follow specific dietary measures for health purposes that conflict with the study diets.
* Use of insulin or sulfonylurea (SU)-derivates.
* Language barrier.
* Pregnancy or lactating.
* Serum potassium > 5.0 mmol/L that requires dietary measures.
* Moderate or severe malnutrition (Patient-Generated Subjective Global Assessment (PG-SGA) stage B or C). In this case, patient will be referred to a renal dietician.
* Participation in other intervention trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  Change in systolic blood pressure (in mmHg)

SECONDARY OUTCOMES:
Cardio-metabolic risk factors (lipids) | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in circulating triglyceride concentrations, low-density lipoprotein cholesterol (LDL-C) and HDL-C (in fasting serum levels) in mmol/L.
Cardio-metabolic risk factors (diastolic blood pressure) | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  Change in diastolic blood pressure (in mmHg)
Cardio-metabolic risk factors (waist circumference) | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in waist circumference (WC) in cm
Cardio-metabolic risk factors (insulin resistance) | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in insulin resistance measuring by the homeostatic model assessment of insulin resistance (HOMA-IR index, fasting glucose, insulin)
Body composition | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in fat and muscle mass measured by multi-frequency bio-electrical impedance analysis (BIA) BMI, weight
Anthropometric measures | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  Change in weight in kilograms
Anthropometric measures II | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  Change in Body Mass Index (BMI) in kilograms per square meter
Body composition II | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in fat and muscle mass measured by multi-frequency bio-electrical impedance analysis (BIA)
Quality of life (QoL) | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in QoL, 12-item short form health survey (SF-12)
Fatigue | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in fatigue (measured by Dutch Checklist Individual Strength (CIS-20) questionnaire)
Physical functioning | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in Hand Grip Strength (HSG)
Physical functioning II | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in the five time sit to stand (FTSTS) test
Nutritional intake | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in nutritional intake measured by a 3-day food diary
Nutritional intake II | before and after experimental diet (high-protein, carbohydrate-reduced diet - 6 weeks) / before and after active comparator (Dutch Nutritional Guidelines - 6 weeks) / wash-out period in between (6 weeks)
  change in nutritional intake measured by nutritional intake biomarkers from 24-hour urine measurements (sodium, potassium, and urea excretion for calculating the protein intake by use of the Maroni equation)

IPD SHARING:
Plan to Share IPD: Undecided